CLINICAL TRIAL: NCT02728128
Title: Platelet and Tissue cAMP: Novel Biomarkers of Milrinone Efficacy in Children
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-2239
Record Dates: First submitted 2016-03-08; First posted 2016-04-05 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Pediatrics; Heart Failure; Congenital Heart Disease; Therapeutics
Keywords: Milrinone
MeSH Terms: conditions — Heart Failure; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urine samples will be retained for future studies once initial analyses have been performed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low cardiac output syndrome: Patients who experience low cardiac output syndrome
- No low cardiac output syndrome: Group that does not experience low cardiac output syndrome.

SUMMARY:
The purpose of this study is to identify if circulating platelet cyclic adenosine monophosphate (cAMP) levels can be used as a biomarker of milrinone efficacy in children following cardiac surgery or undergoing heart transplant.

DETAILED DESCRIPTION:
Milrinone is a phosphodiesterase type III (PDE3) inhibitor with sites of action in cardiac and vascular smooth muscle. PDE3 hydrolyzes the critical second messenger cyclic adenosine monophosphate (cAMP), and PDE3 inhibition (PDE3i) results in a positive inotropic effect in the heart through an increase in cAMP. PDE3i causes relaxation of the vascular smooth muscle and induces vasodilation while concomitantly reducing myocardial oxygen consumption.

In adults, long term PDE3i results in malignant arrhythmias and an increased risk of sudden death, and is therefore not a recommended therapy in this population. However, in the pediatric Heart Failure (HF) population, long-term outpatient milrinone infusions are safely used as a palliative therapy or as a bridge to transplant without an increased risk of unexpected deaths, and results in fewer HF emergency department visits and admissions and improved New York Heart Association (NYHA)/Ross classification. In addition, short term PDE3i (i.e. milrinone) is successfully and routinely used in children presenting with decompensated HF following cardiac surgery. In children undergoing cardiac surgery with cardiopulmonary bypass there is a predictable fall in cardiac index 6 to 18 hours after cardiac surgery. This phenomenon is known as low cardiac output syndrome (LCOS) and is typified by tachycardia and poor perfusion resulting in end-organ dysfunction and risk for cardiac arrest. Milrinone is the only proven drug for prophylactic use in children following cardiac surgery for the prevention of LCOS.

While standard dosing of milrinone is routinely used in children, the actual dose-response relationship is unknown. Indeed, the investigators have noted significant variability in serum milrinone concentrations between patients despite weight based dosing strategies. This uncertainty in dosing is confounded by differences in patient age, size and ontologic maturation of the kidneys. Milrinone dose adjustments, therefore, vary widely among practitioners based on urine output, degree of systemic vasodilation and a change in serum creatinine. Additional uncertainty resides in the inability to easily identify the most appropriate milrinone dose to produce a biological effect (such as an increase in the critical secondary messenger, (cAMP) in the pediatric population.

Because milrinone is excreted as unchanged drug in the urine, kidney function is a critical factor in milrinone dosing. Recently published data demonstrate that 73% of milrinone levels in children with acute kidney injury (AKI) were outside the therapeutic range. Thus, children are particularly vulnerable to inappropriate milrinone dosing. Currently, AKI is diagnosed by an increase in serum creatinine (SCr). Unfortunately, the increase in SCr may not occur until 3 days after AKI occurs. Thus, in children treated with milrinone, undetected AKI would result in significant over-dosing. Since milrinone is also a potent vasodilator, excess milrinone dosing in AKI could lead to hypotension - and further exacerbation of AKI. Therefore, early detection of AKI is especially important in children receiving milrinone. Preliminary data demonstrate that supra therapeutic milrinone concentrations and urinary AKI biomarkers increase in advance of SCr in patients with AKI. In this grant, the investigators propose to determine if increases in Tissue inhibitor metalloproteinase and insulin like growth factor binding protein-7 (TIMP2xIGFBP7) (prior to an increase in SCr) will correlate with increased platelet cAMP and supra-therapeutic milrinone levels.

In the absence of the ability to identify the optimal dose, children are at risk for clinically relevant over or under-dosing with milrinone that can lead to hemodynamic compromise and end organ dysfunction. While clinical response to milrinone remains the most important factor in dose titration decisions, in order to fully optimize milrinone dosing and minimize drug-related toxicity, a biomarker representative of biologic milrinone effect is needed. The Investigators recently demonstrated that milrinone treatment results in increased myocardial cAMP levels and augmented phospholamban phosphorylation in children, but not in adults, with idiopathic dilated cardiomyopathy. In addition, preliminary data suggest that platelet cAMP levels correlate with tissue levels. The purpose of this study is to determine if platelet cAMP levels can serve as a circulating biomarker for end organ (cardiac) milrinone efficacy, and investigate whether changes in this biomarker correlate with clinical efficacy. Defining platelet cAMP levels in pediatric patients with heart disease would provide the basis for a personalized approach to milrinone dose titration and allow identification of those most likely to benefit from its use.

ELIGIBILITY:
Inclusion Criteria:

* Children aged birth to 18 year of age
* Surgical complexity STAT score > 3
* Use of cardiopulmonary bypass for cardiac surgery
* Use of milrinone intra-operatively and post-operatively

Exclusion Criteria:

* Patients on milrinone therapy prior to surgery
* Gestational age less than 34 weeks at the time of surgery
* Weight less than 2500 grams at the time of surgery
* Abnormal renal function prior to cardiac surgery. Abnormal renal function is defined as a serum creatinine > 0.3mg/dL above baseline (lowest value in the preceding 3 months prior to surgery) compared to the level obtained immediately prior to cardiac surgery.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing cardiac surgery with the use of cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Time to the development of low cardiac output syndrome | Within 36 hours following cardiac surgery
  Criteria for low cardiac output

CONTACTS AND LOCATIONS:
Overall Officials: Katja M Gist, DO, MSCS, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DiBianco R, Shabetai R, Kostuk W, Moran J, Schlant RC, Wright R. A comparison of oral milrinone, digoxin, and their combination in the treatment of patients with chronic heart failure. N Engl J Med. 1989 Mar 16;320(11):677-83. doi: 10.1056/NEJM198903163201101. PMID 2646536
- [Background] Ewy GA. Inotropic infusions for chronic congestive heart failure: medical miracles or misguided medicinals? J Am Coll Cardiol. 1999 Feb;33(2):572-5. doi: 10.1016/s0735-1097(98)00596-8. No abstract available. PMID 9973041
- [Background] Hauptman PJ, Mikolajczak P, George A, Mohr CJ, Hoover R, Swindle J, Schnitzler MA. Chronic inotropic therapy in end-stage heart failure. Am Heart J. 2006 Dec;152(6):1096.e1-8. doi: 10.1016/j.ahj.2006.08.003. PMID 17161059
- [Background] Felker GM, O'Connor CM. Inotropic therapy for heart failure: an evidence-based approach. Am Heart J. 2001 Sep;142(3):393-401. doi: 10.1067/mhj.2001.117606. PMID 11526351
- [Background] Nony P, Boissel JP, Lievre M, Leizorovicz A, Haugh MC, Fareh S, de Breyne B. Evaluation of the effect of phosphodiesterase inhibitors on mortality in chronic heart failure patients. A meta-analysis. Eur J Clin Pharmacol. 1994;46(3):191-6. doi: 10.1007/BF00192547. PMID 8070498
- [Background] Packer M, Carver JR, Rodeheffer RJ, Ivanhoe RJ, DiBianco R, Zeldis SM, Hendrix GH, Bommer WJ, Elkayam U, Kukin ML, et al. Effect of oral milrinone on mortality in severe chronic heart failure. The PROMISE Study Research Group. N Engl J Med. 1991 Nov 21;325(21):1468-75. doi: 10.1056/NEJM199111213252103. PMID 1944425
- [Background] Packer M, Medina N, Yushak M. Hemodynamic and clinical limitations of long-term inotropic therapy with amrinone in patients with severe chronic heart failure. Circulation. 1984 Dec;70(6):1038-47. doi: 10.1161/01.cir.70.6.1038. PMID 6388899
- [Background] Price JF, Towbin JA, Dreyer WJ, Moffett BS, Kertesz NJ, Clunie SK, Denfield SW. Outpatient continuous parenteral inotropic therapy as bridge to transplantation in children with advanced heart failure. J Card Fail. 2006 Mar;12(2):139-43. doi: 10.1016/j.cardfail.2005.11.001. PMID 16520263
- [Background] Birnbaum BF, Simpson KE, Boschert TA, Zheng J, Wallendorf MJ, Schechtman K, Canter CE. Intravenous home inotropic use is safe in pediatric patients awaiting transplantation. Circ Heart Fail. 2015 Jan;8(1):64-70. doi: 10.1161/CIRCHEARTFAILURE.114.001528. Epub 2014 Dec 3. PMID 25472966
- [Background] Berg AM, Snell L, Mahle WT. Home inotropic therapy in children. J Heart Lung Transplant. 2007 May;26(5):453-7. doi: 10.1016/j.healun.2007.02.004. PMID 17449413
- [Background] Hoffman TM, Wernovsky G, Atz AM, Bailey JM, Akbary A, Kocsis JF, Nelson DP, Chang AC, Kulik TJ, Spray TL, Wessel DL. Prophylactic intravenous use of milrinone after cardiac operation in pediatrics (PRIMACORP) study. Prophylactic Intravenous Use of Milrinone After Cardiac Operation in Pediatrics. Am Heart J. 2002 Jan;143(1):15-21. doi: 10.1067/mhj.2002.120305. PMID 11773907
- [Background] Gist KM, Mizuno T, Goldstein SL, Vinks A. Retrospective Evaluation of Milrinone Pharmacokinetics in Children With Kidney Injury. Ther Drug Monit. 2015 Dec;37(6):792-6. doi: 10.1097/FTD.0000000000000214. PMID 25860636